CLINICAL TRIAL: NCT01885832
Title: Safety and Feasibility Study of Autologous Stromal Vascular Fraction (SVF) Cells for Treatment of Osteoarthritis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: per sponsor decision
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-SVF-OA-002-2013
Record Dates: First submitted 2013-06-18; First posted 2013-06-25 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Osteoarthritis
Keywords: autologous adipose stem cells; stromal vascular fraction; osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): In the treatment arm, autologous stromal vascular fraction (SVF) will be injected into joints of 20 patients with grade 2, 3, or 4 radiographic OA severity.
  Interventions: Biological: Autologous adipose tissue stromal vascular fraction

INTERVENTIONS:
Biological: Autologous adipose tissue stromal vascular fraction

SUMMARY:
Autologous stromal vascular fraction (SVF) injected into joints of 20 patients with grade 2, 3, or 4 radiographic OA severity will be safe and feasible as assessed by lack of treatment associated adverse events. Improvements in joint function as assessed by Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) are anticipated.

DETAILED DESCRIPTION:
The proposed study is a single center, unblinded, non randomized, phase I/II trial in which the patients will be treated with a single dose of autologous stromal vascular cells (SVF) isolated from 500 ml of adipose tissue extracted from the infraumbilical area. The cellular product will be administered via intra-articular injection into patients with moderate to severe osteoarthritis (OA). Administration will be performed by injection into the synovial space. The dosing regimen will consist of two intraarticular injection of autologous SVF into the index knee. Total injection volume will be about 30 mL in two 15 mL aliquots via a 23 gauge needle inserted 1.5 cm. deep into the intraauricular space of the knee. The total number of SVF to be injected is 1.0 x 10(7) to 5 x 10(7).

The purpose of this study will be to define the safety and efficacy of SVF therapy in improving joint function and the quality of life in patients with OA of the knee. We plan to enroll twenty subjects for treatment for an adequate sample size for safety analysis with signals of efficacy. The primary safety outcome will be tabulation of adverse events related to treatment. Efficacy will be quantified at 3, 6 and 12 months by the total Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).

ELIGIBILITY:
Inclusion Criteria:

Age >18 years and ability to understand the planned treatment.

Idiopathic or secondary osteoarthritis of the knee with grade 2, 3, or 4 radiographic severity, as defined by the modified Kellgren-Lawrence classification

Ability and willingness to undergo liposuction

Exclusion Criteria:

Pregnant women or cognitively impaired adults.

Presence of large meniscal tears ("bucket handle" tears), as detected by clinical examination or by magnetic resonance imaging.

Inflammatory or postinfectious arthritis.

More than 5 degrees of varus or valgus deformity.

Kellgren Lawrence grade 4 osteoarthritis in two compartments (the medial or lateral compartments of the tibiofemoral joint or the patellofemoral compartment) in persons over 60 years of age.

Intraarticular corticosteroid injection within the previous 3 months.

A major neurologic deficit.

Serious medical illness with a life expectancy of less than 1 year.

Prior admission for substance abuse

Body Mass Index (BMI) of 40 kg/m2 or greater

Patient receiving experimental medication or participating in another clinical study within 30 days of signing the informed consent

In the opinion of the investigator or the sponsor the patient is unsuitable for cellular therapy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 6 months

SECONDARY OUTCOMES:
Change from baseline Kellgren-Lawrence classification at 6 months | 6 months
Change from baseline WOMAC Assessment at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Paz-Rodriguez, M.D., Principal Investigator — Stem Cell Institute Panama
Locations (1):
- Stem Cell Instsitute, Panama City, Panama